CLINICAL TRIAL: NCT00770783
Title: Efficacy of Magnetic Seizure Therapy (MST) in Refractory Major Depression
Brief Title: Magnetic Seizure Therapy (MST) for Treatment Resistant Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, MD, Professor of Psychiatry and Psychotherapy, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSG-05-001
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Seizure Therapy (MST) (Experimental)
  Interventions: Device: Tonica MagPro MST
- Electroconvulsive Therapy (ECT) (Active Comparator)
  Interventions: Device: Thymatron

INTERVENTIONS:
Device: Thymatron — Right unilateral placement, 3x seizure threshold, 3 times per week for 4 weeks
  Arms: Electroconvulsive Therapy (ECT)
Device: Tonica MagPro MST — 100% power, vertex placement, 3 times per week for 4 weeks
  Arms: Magnetic Seizure Therapy (MST)

SUMMARY:
The investigators intend to test in a single center, clinical pilot efficacy study the primary hypothesis that Magnetic Seizure Therapy (MST) as add-on therapy to a controlled pharmacotherapy is efficacious in the treatment of refractory major depression assessed with the Hamilton Depression Rating Scale (HAMD).

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with a major depressive episode (MDE) according to DSM-IV Diagnosis Criteria derived from the SCID.
* Patient has not had an acceptable clinical response due to failure (resistance) with at least two treatments from different treatment categories during the current MDE.
* Patient has a score ≥ 20 on the 24-item Hamilton Rating Scale of Depression.
* Patient is able to give his informed consent to participate in this study and he is able to fulfill the requirements of the study.
* Patient is a male or nonpregnant female adequately protected from conception. Females of childbearing potential must use an acceptable method of birth control.
* Convulsive therapy clinically indicated

Exclusion Criteria:

* Patient currently has a secondary diagnosis of, or signs of, delirium, dementia, amnesia, or other cognitive disorders per DSM-IV.
* Patient has had or has currently a diagnosis of non-affective psychotic disorder per DSM-IV.
* Patient has had alcohol or substance dependence within the previous 12 months or abuse within the previous six months other than nicotine dependence or abuse.
* Patient has a history or diagnosis of clinically relevant cardiac disease.
* Patient has a history or diagnosis of clinically relevant injury or disease of the central nervous system.
* Patient has magnetic material in the head.
* Patient has implanted medical devices such as cardiac pacemaker, vagus nerve stimulator, medical pumps etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-02 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clinical improvement (Hamilton Rating Scale for Depression) | After each treatment and at followups up to 3 months after the treatment course

SECONDARY OUTCOMES:
Clinical improvement (Montgomery- Åsberg Rating Scale for Depression) | After each treatment and at followups up to 3 months after the treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Schlaepfer, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- Department of Psychiatry and Psychotherapy - University Hospital, Bonn, Germany

REFERENCES:
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914